CLINICAL TRIAL: NCT04876911
Title: A Single Case Experimental Design Study to Explore the Use of Simulated Presence Therapy as a Formulation Based Intervention for Patients With Dementia Who Are Presenting in Distress.
Brief Title: An Exploration of Simulated Presence Therapy as a Formulation Based Intervention for Dementia Related Distress.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: GN21MH088; 294075 (Other: IRAS)
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Behavioural and Psychiatric Symptoms of Dementia; Stress, Psychological
Keywords: Simulates Presence Therapy; SPT; formulation; electronic device; touchscreen; Intervention; psychosocial; psychological; dementia; dementia care; Newcastle formulation
MeSH Terms: conditions — Stress, Psychological; Dementia

STUDY DESIGN:
Intervention Model Description: Multiple Baseline Single Case Experimental Design (SCED) of two phases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control/Usual Care (No Intervention): No intervention delivered and care is provided as usual.
- Simulated Presence Therapy (SPT) (Experimental): Participants begin to receive the SPT.
  Interventions: Behavioral: Simulated Presence Therapy

INTERVENTIONS:
Behavioral: Simulated Presence Therapy — A video recording of a loved one is played (via an iPad) prior to or during periods where a participant is presenting with stressed/distressed behaviours.
  Other Names: SPT; Simulated Presence Intervention
  Arms: Simulated Presence Therapy (SPT)

SUMMARY:
It is known that persons with a diagnosis of dementia can experience distress associated with the condition. There are different ways that distress is expressed between these persons, but some common occurrences include physical or verbal aggression, tearfulness, upset, confusion and asking repetitive questions. Medications have typically dominated management of symptoms of distress in dementia, and whilst effective, can result in other problems, such as dependency and reduced effectiveness over time. Non-medical interventions may help to reduce distress without the pitfalls of medications. One such intervention is Simulated Presence Therapy.

Simulated Presence Therapy involves playing an audio and/or visual recording with a comforting message from a loved one to a person with dementia to reduce distress. At present, there are few studies examining its effectiveness, with some indication that Simulated Presence Therapy can benefit some people, but this outcome is not consistent. One reason for this may be due to the focus on diagnosis and symptoms in previous studies rather than 'formulation'. Formulation is an approach to healthcare that attempts to arrive at an understanding of a patient's concern(s), taking into account the views of the patient, their loved ones and other healthcare professionals, as well as psychological theory and research evidence.

This study aims to determine if Simulated Presence Therapy delivered via an iPad, when used within a formulation, reduces distress in patients with moderate to severe dementia admitted for long-term care in a care home or inpatient hospital ward. This study will also examine how user-friendly and helpful Simulated Presence Therapy was for healthcare professionals who administer it. Participants may not have the ability to provide consent; therefore, this will be obtained from the legal guardian or next of kin.

All participants will have received a formulation that identifies Simulated Presence Therapy as the preferred intervention. Their occurrence will be counted on a chart and tallied each day before and after the intervention is introduced. The healthcare staff who administer Simulated Presence Therapy will complete a questionnaire to evaluate their opinions on its user-friendliness and effectiveness. It is hoped that this study may enable service providers to better understand how to integrate Simulated Presence Therapy into healthcare services for persons with a diagnosis of dementia.

DETAILED DESCRIPTION:
Background: Persons with dementia (PwD) often present with a cluster of signs or symptoms of distorted perceptions, thoughts, mood and behaviours, commonly referred to as the behavioural and psychological symptoms of dementia. Psychosocial conceptualisations posit that these symptoms manifest as a result of distress arising from an unmet need; thus, the term 'stressed and distressed behaviours' (SDB) may more accurately represent the aetiology of these symptoms. This ethos has been aggregated into the Newcastle model, first conceptualised by Dr Ian James and his colleagues, which emphasises a formulation-based approach to dementia care. Formulation refers to the process of collaboratively developing a hypothesis regarding an individual's difficulties by incorporating psychological theory and evidence.

Although formulation-based approaches are become more widespread, prescribing practices for medical treatments remains suboptimal across dementia care settings. Considering the personal, societal and economic burdens of SDB in PwD, coupled with the disadvantages of pharmacological interventions, there remains a real need to develop effective non-pharmacological, psychosocial alternatives. One such intervention is Simulated Presence Therapy (SPT).

SPT is an intervention that involves playing a video and/or audio recording of a loved one to a PwD with a reassuring message when they present with SDB. Studies examining the efficacy of SPT are sparse; however, what little research that has been conducted has highlighted its effectiveness in some instances. Thus far, studies have not explored SPT when it has been identified as a way of addressing an unmet need through a formulation-driven assessment process. Instead, it has been applied to participants within specific care settings with a symptom rather than formulation-based approach. Hence, this study will explore the efficacy of SPT as part of a formulation-driven approach, grounded in the Newcastle model.

Aim/objectives (s): The present study will aim to investigate the efficacy of SPT for SDB in PwD when it has been specifically identified via a Newcastle formulation as the preferred intervention within care homes and hospital wards operated by the National Health Service of Greater Glasgow and Clyde (NHSGGC) and their associated Health and Social Care Partnerships (HSCP). The research is being conducted to fulfil part of the requirements of the Principal Investigator's Doctorate in Clinical Psychology Qualification at the University of Glasgow, and the University will therefore be an additional collaborating organisation. In terms of objectives:

* Primary Objective - Introduction of SPT will significantly reduce SDB during day-to-day activities when compared to activities without SPT.
* Secondary Objective - What is the acceptability of SPT amongst healthcare professionals that administer it?

Design: This study will employ a randomised single case experimental design (SCED) of two phases (i.e. AB) with multiple baselines. This which would involve randomly allocating PwD to a staggered baseline period (A), followed by the intervention phase (B), which would last as long as the corresponding baseline phase.

Sample: Owing to the fact that, whilst the PwD are the participants that will form the key group to answer the research question, from a technical perspective, the sample consists of multiple categories of persons. For clarity, the following terms are employed:

1. 'Participants' will refer to the PwD recruited to receive SPT.
2. 'Informants' will refer to the person who complete the two attachment/relationship questionnaires for the participant.
3. 'Recorders' will refer to non-healthcare professionals, such as family members or friends, who agree to be filmed for the SPT video.
4. 'Professionals' will refer to the care staff involved in the PwD's care who complete the staff user-experience questionnaire within this study.
5. 'Sample' will refer to all persons participating in the study (i.e. Participants, Informants, Recorders and Professionals).

The anticipated minimum sample size is 13, consisting of participants (N = 6), informants/recorders (N = 6) and professional(s) (N = 1). Recruitment will be from identified care homes and hospital wards that receive input from NHSGGC's Older Person Psychology Service (OPPS).

Measure(s):

* Dementia Severity Rating Scale (DSRS) - This is a validated multiple-choice, informant-based questionnaire, designed to categorise the severity of a patient's dementia. These categories are 'mild', 'moderate' or 'severe'.
* Measure of Attachment Adapted (MOA) - This is a measure of attachment that has been adapted by the Principal Investigator for use in the present study and to be answered by informants. Informants are asked to read three paragraphs and asked to tick which one they feel best describes the patient. There are two sections of the measure: (1) One for if the informant has known the patient before they received their diagnosis of dementia, and (2) another for if the informant knew the patient ONLY after they received a diagnosis. The informant needs to only complete one of these sections. Attachment style can then be categorised as 'secure', 'avoidant' or 'anxious/ambivalent'.
* Measure of Attachment Qualities Adapted (MAQ) - This is a multiple-choice, Likert-scale measure of attachment that has been adapted by the Principal Investigator for use in the present study and to be answered by informants. There are two sections of the measure: (1) One for if the informant has known the patient before they received their diagnosis of dementia, and (2) another for if the informant knew the patient ONLY after they received a diagnosis. The informant needs to only complete one of these sections. Attachment style can then be categorised as 'secure', 'avoidant', 'ambivalent-worry' or 'ambivalent-merger'.
* Unified Theory of Acceptance and Use of Technology (UTAT)-informed Questionnaire - This is a self-report, Likert scale questionnaire developed by the Principal Investigator based on the UTAT. The measure consists of a series of statements pertaining to the usefulness and effectiveness of SPT with respondents who administered SPT selecting how strongly they agree/disagree with each. Higher scores are indicative of greater usefulness, acceptability and/or effectiveness.
* Frequency Chart - This is a chart which is used to tally the number of dSDB exhibited by patients within a specific time period and day. These recordings are made by healthcare staff who work directly with a patient.

Procedures: The process for recruitment is as follows: where capacity to consent is retained, this will be sought from the participant; where the participant is deemed to not have capacity to consent, informed consent for will be obtained from the relevant legal guardian/next of kin; informed consent for those persons who are not healthcare professionals, but complete questionnaires and record videos for the participants, will also be obtained with regard to inclusion of their responses within the present study. Informed consent for the staff UTAT-informed questionnaire will also be obtained.

Following the recruitment process, arrangements to obtain recordings and complete the MOA and MAQ will be established collaboratively between the person recorded and NHSGGC OPPS. All participants will have already received a Newcastle formulation as part of routine care and will be randomly allocated to randomly allocated to a 14, 17 or 21-day baseline period where dSDB is tallied. Immediately once the baseline phase has concluded, the intervention phase will commence, which will last indefinitely for the participants for whom SPT is an effective intervention, although the data that will be extracted at intervention stage will be at least the length of the baseline.

The UTAT-informed questionnaire would be disseminated to professionals near the conclusion of the data collection stage.

Data Analysis: Data analysis for evaluating intervention effects in SCEDs encompasses visual inspection and statistical analysis. Visual analysis involves examining level, trend, variability, immediacy of effect, overlap, and consistency of data patterns within and between phases. Statistical analysis will involve calculation of a Baseline Corrected Tau (BC-Tau) to measure data non-overlap between the two phases (A and B). Non-overlapping data as an indicator of performance difference between phases is included in standards for evaluating SCEDs. Additionally, BC-Tau is useful in aggregating data across phases to produce an overall effect size.

Evaluation of the secondary objective will involve calculating the average score across participants on the UTAT informed questionnaire, with a higher score indicative of greater acceptability.

Ethics and safety: A number of safeguards are in place regarding sample and researcher safety with relevant policies and legislation consulted in the construction of this project. These are detailed in full within the uploaded research protocol. Applications/approvals will be sought by an Ethics committee and NHSGGC's Research and Innovation department. Approval to proceed to ethics for this project has been obtained from the University of Glasgow.

Timetable:

* May/June 2021: Ethics submission.
* June/July 2021 - December 2021: Recruitment and data collection.
* January 2022: End of data collection, data analysis and write-up.
* February-April 2022: Final report article generated.

Dissemination/application: The results of this study will provide insight into the efficacy of SPT when used as part of a formulation-driven approach to dementia care. It is anticipated that this information will enable service providers to understand how to integrate SPT in services and care pathways for PwD. Dissemination will occur once the final research article has been generated by the Principal Investigator, which will be made available on the University of Glasgow's Enlighten thesis repository for public domain access in PDF format, and possibly in a paper that will be submitted for publication.

ELIGIBILITY:
Inclusion Criteria:

For participants:

* A resident within a care home or hospital ward setting operated by NHS Greater Glasgow and Clyde and/or Glasgow City HSCP, Inverclyde HSCP and/or Renfrewshire HSCP.
* Persons aged ≥ 65 years.
* First language must be English.
* A diagnosis of any form of dementia within the moderate to severe stages, defined as a score of at least '19' on the validated Dementia Severity Rating Scale.
* Present with SDB as confirmed by a Newcastle formulation constructed by a psychologist with multidisciplinary input.
* Having retained the relevant cognitive faculties required to engage with audio-video technologies, including attention, recognition and communication as confirmed by a Newcastle formulation constructed by a clinical psychologist with multidisciplinary input.

For informants, inclusion requires proficiency in the English language and having known the participant before and/or after the participants diagnosis of dementia, as well as having interacted with the participant in any capacity over the previous year.

For recorders, inclusion criteria involved proficiency in English language and ongoing contact/interaction with the participant for whom the recording is being made. This would be made clear through consultation with the care team and the Newcastle formulation that will have been made as part of routine practice.

Finally, regarding professionals, inclusion involves proficiency in English language and being employed by NHSGGC and having worked directly on a regular basis with the participant at point of recruitment (i.e. once over the previous 3-month period).

Exclusion Criteria:

For participants:

* No relative/friend/caregiver available to be recorded.
* Significant vision and/or hearing impairments that cannot be corrected.
* Pre-existing neurological or severe psychiatric disorder (e.g. psychosis, bi-polar disorder).
* Diagnosed or suspected intellectual and developmental disability.

For informants, the main exclusion criteria include being unable to understand English.

For the recorders, exclusion criteria involve possible speech deficits or issues that may impact the quality of the recording and/or having a full face covering that prevents a recognition of a person on video. Additionally, if someone does not have a close relationship or has a contentious relationship with the participant, they would not be eligible to be recorded. This would be made clear through consultation with the care team and the Newcastle formulation that will have been made by the team as part of routine practice.

Finally, regarding professionals, the main exclusion criteria would be not having been familiarised with the SPT procedure.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Frequency Chart | 21 to 48 days
  A frequency chart which is used to tally the occurrence of stressed/distressed behaviours per day by healthcare staff.

SECONDARY OUTCOMES:
UTAT-informed staff questionnaire | 10-15 minuted per participant.
  Self-report questionnaire developed by the Principal Investigator to ascertain how user-friendly and effective SPT was for healthcare staff who employed it.

CONTACTS AND LOCATIONS:
Overall Officials: Danyal A Ansari, BA, MSc, Principal Investigator — NHSGGC and University of Glasgow
Locations (1):
- NHSGGC, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This project forms part of a thesis and IPD would not be shared with others.

REFERENCES:
- [Background] Abraha I, Rimland JM, Lozano-Montoya I, Dell'Aquila G, Velez-Diaz-Pallares M, Trotta FM, Cruz-Jentoft AJ, Cherubini A. Simulated presence therapy for dementia. Cochrane Database Syst Rev. 2017 Apr 18;4(4):CD011882. doi: 10.1002/14651858.CD011882.pub2. PMID 28418586
- [Background] Carver, C. S. (1997). Adult attachment and personality: Converging evidence and a new measure. Personality and Social Psychology Bulletin, 23(8), 865-883. https://doi.org/10.1177/0146167297238007
- [Background] Clark CM, Ewbank DC. Performance of the dementia severity rating scale: a caregiver questionnaire for rating severity in Alzheimer disease. Alzheimer Dis Assoc Disord. 1996 Spring;10(1):31-9. PMID 8919494
- [Background] Hazan C, Shaver P. Romantic love conceptualized as an attachment process. J Pers Soc Psychol. 1987 Mar;52(3):511-24. doi: 10.1037//0022-3514.52.3.511. PMID 3572722
- [Background] James, I. A. (2011). Understanding behaviours in dementia that challenge. Jessica Kingsley Publishers.
- [Background] Tible OP, Riese F, Savaskan E, von Gunten A. Best practice in the management of behavioural and psychological symptoms of dementia. Ther Adv Neurol Disord. 2017 Aug;10(8):297-309. doi: 10.1177/1756285617712979. Epub 2017 Jun 19. PMID 28781611
- [Background] Venkatesh, V., Morris, M. G., Davis, G. B., & Davis, F. D. (2003). User acceptance of information technology: Toward a unified view. MIS Quarterly: Management Information Systems, 27(3), 425-478. https://doi.org/10.2307/30036540